CLINICAL TRIAL: NCT07249762
Title: Surgical Critical Care Initiative (SC2i) Tissue and Data Acquisition Protocol (TDAP) in Burn Patients Improving the Robustness and Generalizability of Post-burn Sepsis Prediction With the Post-Burn Sepsis Digital Twin. Group 1
Status: Not yet recruiting | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Emory University (Other); United States Army Institute of Surgical Research (U.S. Federal Agency); University of South Florida (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: USUHS.2025-153; HT94252320022 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Burn Injury; Wound Healing; Critical Illness; Multiple Organ Dysfunction Syndrome
Keywords: Burn Infection; Sepsis; Critical Illness; Thermal Injury; Infection; Multiple Organ Dysfunction Syndrome (MODS); Acute Respiratory Distress Syndrome (ARDS); Wound Healing; Biomarkers; Digital Twin Model; Predictive Analytics; Surgical Critical Care
MeSH Terms: conditions — Sepsis; Burns; Critical Illness; Multiple Organ Failure; Infections; Respiratory Distress Syndrome | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During this study, small amounts of blood will be collected from participants at scheduled times. Whenever possible, these samples will be taken during routine blood draws to avoid extra needle sticks. The total amount of blood collected for research will be limited to safe levels. If participants need surgery to remove damaged skin, small pieces of tissue that would normally be thrown away may also be saved for research. These samples will be used to study how the body responds to burn injury and recovery. All samples will be labeled with a study code only, not personal identifiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1 - Minimal Risk Burn Patient: The study includes adult patients (18 years and older) admitted with significant burn injuries involving more than 10% of their total body surface area (TBSA) who require surgical management and/or care within a surgical critical care setting. As part of their participation, small amounts of blood are collected at scheduled times during hospitalization, and small pieces of skin or tissue normally removed during burn surgery may also be saved. Medical information already recorded in the hospital chart-such as vital signs, lab results, surgeries, and complications-is also included in the study.
  Interventions: Other: Observational Cohort (No Intervention)

INTERVENTIONS:
Other: Observational Cohort (No Intervention) — This is not a treatment trial-no drugs, devices, or procedures are being tested. Participants receive standard burn care only. The research involves collecting blood and tissue samples (when clinically indicated) and reviewing medical record data.
  Other Names: observational

SUMMARY:
This study is following adult patients with serious burn injuries to better understand how their bodies respond to treatment and recovery. Researchers will collect small amounts of blood and tissue samples, along with information already recorded in the medical record, such as vital signs, lab results, and details of surgeries or complications. The goal is to identify patterns that may help predict who is at higher risk for infections or other problems after a burn injury. This information could lead to new tools, including computer-based models, to improve burn care and outcomes in the future. Participation involves providing samples and allowing researchers to review medical records during the hospital stay and up to one year after discharge.

DETAILED DESCRIPTION:
This is a prospective observational study of adult patients with significant burn injuries. The purpose is to understand the body responses to significant burns, treatment, and recovery and to identify factors that predict complications like infection or sepsis. By studying patterns in clinical information, blood, and tissue samples to develop computer-based models intended to improve diagnosis and guide future treatments.

Eligible participants are males and females between 18 and 80 years old with burn injuries involving more than 10% of their total body surface area (TBSA) who require care in a critical care or emergency setting at an SC2i-member facility (e.g., Emory, Grady, USF, USAISR). All participants or their Legally Authorized Representatives (LARs) must provide informed consent. About 40 patients are expected to participate.

ELIGIBILITY:
Inclusion Criteria:

* Burn Injury >10% TBSA with who have a recognized concurrent or impending risk for clinical decompensation.
* Male and female ages 18 years and older (maximum age of 80 years old) with burn injury or related illness requiring surgical care or treatment in a critical care or emergency setting who are being cared for at an SC2i-member clinical care facility (Emory/Grady, USF and USAISR) will be considered for study.
* Ability to understand the purposes and risks of the study and to provide informed consent, either through written documentation or in accordance with the IRB-approved Waiver of Documentation of Consent procedures. In the case of incapacitated patients, a willing Legally Authorized Representative (LAR) may provide informed consent in accordance with written documentation or under the provisions of the approved Waiver of Documentation of Consent.

Exclusion Criteria:

* Any condition that, in the opinion of the attending physician, would place the patient or volunteer subject at undue risk by participating. Specific conditions include but are not limited to anemia prohibitive of phlebotomy, or technical considerations that would prevent acquisition of sufficient tissue for clinical use.
* Pregnant patients
* Minors < 18 years of age
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study of patients with burn wounds >10% TBSA requiring surgical management and/or management within a surgical critical care setting.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Sepsis and Other Major Complications After Burn Injury | During hospitalization, up to 12 months after discharge
  Clinical data will be collected from medical records to capture whether patients develop sepsis, organ dysfunction, or other serious complications following burn injury.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of South Florida - Tampa General Hospital, Tampa, Florida
  - Emory University-Grady Memorial Hospital, Atlanta, Georgia
  - United States Army Institute of Surgical Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including clinical information and research sample data, may be shared with qualified researchers. Data will be stripped of direct identifiers, and a coded study ID will be used. The code key will remain at the enrolling site and will not be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified IPD will be available after primary analyses are complete and results are published, typically within 12-24 months after final data collection.
Access Criteria: Data requests will be reviewed by the study steering committee. Investigators will be required to submit a data use agreement and provide documentation of institutional review/ethics oversight.

REFERENCES:
- [Background] Yan J, Hill WF, Rehou S, Pinto R, Shahrokhi S, Jeschke MG. Sepsis criteria versus clinical diagnosis of sepsis in burn patients: A validation of current sepsis scores. Surgery. 2018 Dec;164(6):1241-1245. doi: 10.1016/j.surg.2018.05.053. Epub 2018 Jul 23. PMID 30049483
- [Background] Boehm D, Menke H. Sepsis in Burns-Lessons Learnt from Developments in the Management of Septic Shock. Medicina (Kaunas). 2021 Dec 24;58(1):26. doi: 10.3390/medicina58010026. PMID 35056334
- [Background] Hampson P, Dinsdale RJ, Wearn CM, Bamford AL, Bishop JRB, Hazeldine J, Moiemen NS, Harrison P, Lord JM. Neutrophil Dysfunction, Immature Granulocytes, and Cell-free DNA are Early Biomarkers of Sepsis in Burn-injured Patients: A Prospective Observational Cohort Study. Ann Surg. 2017 Jun;265(6):1241-1249. doi: 10.1097/SLA.0000000000001807. PMID 27232244
- [Background] Moins-Teisserenc H, Cordeiro DJ, Audigier V, Ressaire Q, Benyamina M, Lambert J, Maki G, Homyrda L, Toubert A, Legrand M. Severe Altered Immune Status After Burn Injury Is Associated With Bacterial Infection and Septic Shock. Front Immunol. 2021 Mar 2;12:586195. doi: 10.3389/fimmu.2021.586195. eCollection 2021. PMID 33737924
- [Background] Sadeq F, Poster J, Chu C, Weber J, Lydon M, Begis MD, Sheridan RL, Uygun K. Specific patterns of vital sign fluctuations predict infection and enable sepsis diagnosis in pediatric burn patients. PLoS One. 2022 Feb 7;17(2):e0263421. doi: 10.1371/journal.pone.0263421. eCollection 2022. PMID 35130306
- [Background] Niggemann P, Rittirsch D, Buehler PK, Schweizer R, Giovanoli P, Reding T, Graf R, Plock JA, Klein HJ. Incidence and Time Point of Sepsis Detection as Related to Different Sepsis Definitions in Severely Burned Patients and Their Accompanying Time Course of Pro-Inflammatory Biomarkers. J Pers Med. 2021 Jul 23;11(8):701. doi: 10.3390/jpm11080701. PMID 34442346
- [Background] Adams R, Henry KE, Sridharan A, Soleimani H, Zhan A, Rawat N, Johnson L, Hager DN, Cosgrove SE, Markowski A, Klein EY, Chen ES, Saheed MO, Henley M, Miranda S, Houston K, Linton RC, Ahluwalia AR, Wu AW, Saria S. Prospective, multi-site study of patient outcomes after implementation of the TREWS machine learning-based early warning system for sepsis. Nat Med. 2022 Jul;28(7):1455-1460. doi: 10.1038/s41591-022-01894-0. Epub 2022 Jul 21. PMID 35864252
- [Background] Henry KE, Adams R, Parent C, Soleimani H, Sridharan A, Johnson L, Hager DN, Cosgrove SE, Markowski A, Klein EY, Chen ES, Saheed MO, Henley M, Miranda S, Houston K, Linton RC 2nd, Ahluwalia AR, Wu AW, Saria S. Factors driving provider adoption of the TREWS machine learning-based early warning system and its effects on sepsis treatment timing. Nat Med. 2022 Jul;28(7):1447-1454. doi: 10.1038/s41591-022-01895-z. Epub 2022 Jul 21. PMID 35864251
- [Background] Tran NK, Albahra S, Pham TN, Holmes JH 4th, Greenhalgh D, Palmieri TL, Wajda J, Rashidi HH. Novel application of an automated-machine learning development tool for predicting burn sepsis: proof of concept. Sci Rep. 2020 Jul 23;10(1):12354. doi: 10.1038/s41598-020-69433-w. PMID 32704168
- [Background] Rashidi HH, Sen S, Palmieri TL, Blackmon T, Wajda J, Tran NK. Early Recognition of Burn- and Trauma-Related Acute Kidney Injury: A Pilot Comparison of Machine Learning Techniques. Sci Rep. 2020 Jan 14;10(1):205. doi: 10.1038/s41598-019-57083-6. PMID 31937795
- [Background] von Lilienfeld-Toal M, Dietrich MP, Glasmacher A, Lehmann L, Breig P, Hahn C, Schmidt-Wolf IG, Marklein G, Schroeder S, Stuber F. Markers of bacteremia in febrile neutropenic patients with hematological malignancies: procalcitonin and IL-6 are more reliable than C-reactive protein. Eur J Clin Microbiol Infect Dis. 2004 Jul;23(7):539-44. doi: 10.1007/s10096-004-1156-y. Epub 2004 Jun 22. PMID 15221617